CLINICAL TRIAL: NCT00719043
Title: A Trial to Evaluate the Safety and Immunogenicity of Monovalent H5N1 Vaccine in Adults >=18 Yrs of Age
Brief Title: Immunogenicity & Safety of GSK's Avian Flu Vaccine 1557484A Given to Adults Aged ≥18 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110624
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: Influenza; H5N1; Avian; Vaccines; Safety; Immunogenicity; Pandemic; Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- A/Indonesia primed-A/turkey Influenza (H5N1)-F1-Placebo Group (Experimental): Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) formulation 1 at Day 0 followed by one booster dose of A/turkey H5N1 vaccine formulation 1 at Day 182 and one dose of placebo (phosphate buffered saline, PBS) at Day 549. Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) and Placebo vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, A/turkey H5N1 vaccine was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia); Biological: Placebo
- A/Indonesia primed-A/turkey Influenza (H5N1)-F2-Placebo Group (Experimental): Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) formulation 2 at Day 0 followed by one booster dose of A/turkey H5N1 vaccine formulation 2 at Day 182 and one dose of placebo (phosphate buffered saline, PBS) at Day 549. Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) and Placebo vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, A/turkey H5N1 vaccine was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia); Biological: Placebo
- A/Indonesia primed-A/turkey Influenza (H5N1)-F3-Placebo Group (Experimental): Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) formulation 3 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 3 at Day 549. Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia); Biological: Placebo
- A/Indonesia primed-Placebo-A/turkey Influenza (H5N1)-F1-Group (Experimental): Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) vaccine formulation 1 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 1 at Day 549. Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia); Biological: Placebo
- A/Indonesia primed-Placebo-A/turkey Influenza (H5N1)-F4-Group (Experimental): Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) formulation 4 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 4 at Day 549. Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia); Biological: Placebo
- A/Indonesia primed-Placebo-A/turkey Influenza (H5N1)-F2-Group (Experimental): Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) formulation 2 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 2 at Day 549. Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia); Biological: Placebo
- Naïve Placebo-A/turkey Influenza (H5N1)-F3-Group (Placebo Comparator): Healthy subjects aged 18 years of age or older at the time of vaccination received one dose of placebo (phosphate buffered saline, PBS) at Day 0 followed by two doses of A/turkey H5N1 vaccine formulation 3, one dose administered at Day 182 and the other at Day 549. Placebo vaccine and one dose of A/turkey H5N1 vaccine (Day 549) was administered intramuscularly in the deltoid region of the non-dominant arm while the other dose of A/turkey H5N1 vaccine (Day 182) was administered intramuscularly in the deltoid region of the dominant arm.
  Interventions: Biological: A/turkey H5N1 vaccine; Biological: Placebo

INTERVENTIONS:
Biological: A/turkey H5N1 vaccine — Administered as an intramuscular (IM) injection
Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted (A/Indonesia) — Administered as an intramuscular (IM) injection
  Arms: A/Indonesia primed-A/turkey Influenza (H5N1)-F1-Placebo Group; A/Indonesia primed-A/turkey Influenza (H5N1)-F2-Placebo Group; A/Indonesia primed-A/turkey Influenza (H5N1)-F3-Placebo Group; A/Indonesia primed-Placebo-A/turkey Influenza (H5N1)-F1-Group; A/Indonesia primed-Placebo-A/turkey Influenza (H5N1)-F2-Group; A/Indonesia primed-Placebo-A/turkey Influenza (H5N1)-F4-Group
Biological: Placebo — Administered as an intramuscular (IM) injection

SUMMARY:
The purpose of this study is to determine whether GSK's avian flu vaccine GSK 1557484A is immunogenic and safe when given to adults aged >=18 years.

This Protocol Posting has been updated following Amendments 1-3 of the Protocol, Dec 2009. The impacted sections are study design and outcome measures.

DETAILED DESCRIPTION:
All subjects will receive 3 doses of study vaccine, including 2 doses of active vaccine and 1 dose of placebo. All subjects will attend formal study center visits for safety and immunogenicity assessments on Days 0, 10, 42, 182, 192, 224, 549, 559, 591, and 729. A telephone contact to assess safety will be made at Day 364 and Day 909.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18 years of age or older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Stable health status as defined by absence of a health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within 1 month prior to enrollment.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
* Subjects who the investigator believes can and will comply with the requirements of the protocol

Exclusion Criteria:

* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Diagnosed with cancer, or treatment for cancer, within 3 years.

  * Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
  * Persons with a history of histologically-confirmed basal cell carcinoma of the skin successfully treated with local excision only are excepted and may enroll within 3 years of diagnosis, but other histologic types of skin cancer require a 3 year untreated and disease-free window as above.
  * Women who are disease-free 3 years or more after treatment for breast cancer and receiving long-term prophylactic tamoxifen are excepted and may enroll.
* Presence of an oral temperature ≥ 37.8ºC, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids (prednisone >= 10 mg/day for more than 14 consecutive days) within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Administration of any vaccines within 30 days before the first study vaccine dose.
* Previous administration of any H5N1 vaccine.
* Use of any investigational or non-registered product (drug or vaccine) or planned participation in another investigational study within 30 days prior to study enrollment, or during the 18 months following the first test article dose. Use of any investigational or non-registered product with immunosuppressive properties is exclusionary at any time during the trial.
* Receipt of any immunoglobulins and/or any blood products within 6 months of study enrollment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins or mercurial preservatives); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result prior to vaccination.
* Lactating or nursing.
* Women of child bearing potential who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to treatments.
* Known receipt of analgesic or antipyretic medication with the specific intent of prophylaxis of vaccine reactogenicity on the day of first or any treatment. Subjects on stable chronic regimens of potentially analgesic or anti-pyretic medications for pre-existing diagnoses are not required to discontinue them (to do so would represent evaluation of combined vaccine reactogenicity AND treatment withdrawal - which is not the intent of the protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2008-07-11; Primary Completion 2010-04-22 (Actual); Study Completion 2011-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (10):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
- Canada (3):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 110624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110624 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study duration was of approximately 909 days for all subjects.
Period: Overall Study
Arm/Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F1-Placebo Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F2-Placebo Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group | Naïve Placebo-A/Turkey Influenza (H5N1)-F3-Group
Started | 120 | 121 | 119 | 119 | 122 | 120 | 120
Completed | 88 (Up to Day 909) | 96 (Up to Day 909) | 99 (Up to Day 909) | 96 (Up to Day 909) | 95 (Up to Day 909) | 86 (Up to Day 909) | 92 (Up to Day 909)
Not Completed | 32 | 25 | 20 | 23 | 27 | 34 | 28
Not completed — Adverse Event | 5 | 1 | 2 | 2 | 1 | 4 | 4
Not completed — Lost to Follow-up | 14 | 10 | 8 | 9 | 10 | 9 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 1 | 2 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 12 | 14 | 9 | 10 | 16 | 18 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F1-Placebo Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F2-Placebo Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group | Naïve Placebo-A/Turkey Influenza (H5N1)-F3-Group | Total
Number analyzed (Participants) | 120 | 121 | 119 | 119 | 122 | 120 | 120 | 841
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (18.01) | 49.6 (17.93) | 50.7 (17.67) | 49.2 (17.75) | 50.3 (17.77) | 50.1 (18.92) | 50.0 (18.03) | 49.95 (17.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 73 | 69 | 70 | 68 | 70 | 75 | 505
  Male | 40 | 48 | 50 | 49 | 54 | 50 | 45 | 336

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. Pre-vaccination for this outcome measure corresponds to Day 549. This outcome concerns solely subjects in the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4 and Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 groups.
Time Frame: At Day 559
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, i.e., all evaluable subjects with at least Day 182 and 192 or Day 549 and 559 haemagglutination inhibition (HI) titer results for the A/turkey/Turkey/1/05 virus.
Measure: Number; unit: Subjects
Arm/Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group
Number analyzed (Participants) | 83 | 87 | 80 | 72
Subjects | 71 | 81 | 73 | 65

2. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. Pre-vaccination for this outcome measure corresponds to Day 182. This outcome concerns solely subjects in the Naïve Placebo-A/turkey H5N1-Formulation 3 Group
Time Frame: At Day 192
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Naïve Placebo-A/Turkey Influenza (H5N1)-F3-Group
Number analyzed (Participants) | 99
Subjects | 44

3. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey) Strain.
Description: HI antibody titers against the A/turkey virus strain were expressed as geometric mean titers (GMTs). This outcome concerns solely subjects in the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4 and Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 groups.
Time Frame: At Days 549 and 559
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group
Number analyzed (Participants) | 83 | 88 | 81 | 72
Titers
  A/turkey, Day 549 (N=83,88,81,72) | 11.1 [8.8 to 14.1] | 8.3 [7.0 to 9.7] | 9.2 [7.6 to 11.2] | 11.4 [9.1 to 14.4]
  A/turkey, Day 559 (N= 83,88,81,72) | 356.7 [265.9 to 478.5] | 266.4 [202.2 to 351.2] | 446.6 [336.0 to 593.7] | 343.9 [254.2 to 465.3]

4. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey) Strain.
Description: HI antibody titers against the A/turkey virus strain were expressed as geometric mean titers (GMTs). This outcome concerns solely subjects in the Naïve Placebo-A/turkey H5N1-Formulation 3 Group.
Time Frame: At Days 182 and 192
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Naïve Placebo-A/Turkey Influenza (H5N1)-F3-Group
Number analyzed (Participants) | 100
Titers
  A/turkey strain, Day 182 (N=100) | 10.8 [8.4 to 13.9]
  A/turkey strain, Day 192 (N=99) | 43.5 [32.6 to 58.0]

5. Primary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome concerns solely subjects in the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4 and Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 groups.
Time Frame: At Days 549 and 559
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group
Number analyzed (Participants) | 88 | 87 | 81 | 72
Subjects
  A/turkey, Day 549 (N=83,88,81,72) | 15 | 8 | 10 | 13
  A/turkey, Day 559 (N= 83,87,80,72) | 79 | 83 | 77 | 69

6. Primary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome concerns solely subjects in the Naïve Placebo-A/turkey H5N1-Formulation 3 Group.
Time Frame: At Days 182 and 192
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Naïve Placebo-A/Turkey Influenza (H5N1)-F3-Group
Number analyzed (Participants) | 100
Subjects
  A/turkey strain, Day 182 (N=100) | 24
  A/turkey strain, Day 192 (N=99) | 64

7. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any was defined as an occurrence of the specified solicited local symptom regardless of its intensity.
Time Frame: Within the 7-day (Days 0-6) post vaccination periods
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one dose of vaccine for whom any post-vaccination data were available.
Measure: Number; unit: Subjects
Groups:
- Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group: Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Pumarix™ vaccine formulation 1 at Day 0 followed by one booster dose of A/turkey H5N1 vaccine formulation 1 at Day 182 and one dose of placebo (phosphate buffered saline, PBS) at Day 549. Pumarix™ and Placebo vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, A/turkey H5N1 vaccine was administered intramuscularly in the deltoid region of the dominant arm.
- Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group: Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Pumarix™ vaccine formulation 2 at Day 0 followed by one booster dose of A/turkey H5N1 vaccine formulation 2 at Day 182 and one dose of placebo (phosphate buffered saline, PBS) at Day 549. Pumarix™ and Placebo vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, A/turkey H5N1 vaccine was administered intramuscularly in the deltoid region of the dominant arm.
- Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group: Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Pumarix™ vaccine formulation 3 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 3 at Day 549. Pumarix™ and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
- Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group: Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Pumarix™ vaccine formulation 1 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 1 at Day 549. Pumarix™ and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
- Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group: Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Pumarix™ vaccine formulation 4 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 4 at Day 549. Pumarix™ and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
- Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group: Healthy subjects aged 18 years of age or older at the time of enrolment were primed with one dose of Pumarix™ vaccine formulation 2 at Day 0, one dose of placebo (phosphate buffered saline, PBS) at Day 182 followed by one booster dose of A/turkey H5N1 vaccine formulation 2 at Day 549. Pumarix™ and A/turkey H5N1 vaccines were administered intramuscularly in the deltoid region of the non-dominant arm while, Placebo vaccine was administered intramuscularly in the deltoid region of the dominant arm.
- Naïve Placebo-A/Turkey H5N1-Formulation 3 Group: Healthy subjects aged 18 years of age or older at the time of vaccination received one dose of placebo (phosphate buffered saline, PBS) at Day 0 followed by two doses of A/turkey H5N1 vaccine formulation 3, one dose administered at Day 182 and the other at Day 549.Placebo vaccine and one dose of A/turkey H5N1 vaccine (Day 549) was administered intramuscularly in the deltoid region of the non-dominant arm while the other dose of A/turkey H5N1 vaccine (Day 182) was administered intramuscularly in the deltoid region of the dominant arm.
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 120 | 121 | 119 | 119 | 122 | 120 | 120
Subjects
  Any Pain | 98 | 100 | 101 | 93 | 102 | 90 | 95
  Any Redness | 8 | 4 | 12 | 9 | 14 | 4 | 8
  Any Swelling | 6 | 7 | 15 | 4 | 16 | 9 | 11

8. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, headache, joint pain at other locations (joint pain), muscle aches, shivering, sweating and fever. Any was defined as an occurrence of the specified solicited general symptom, irrespective of its intensity or relationship to vaccination. Any fever was defined as oral temperature higher than or equal to (≥) 38.0 degrees Celsius (°C).
Time Frame: Within the 7-day (Days 0-6) post vaccination periods
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 120 | 121 | 119 | 119 | 122 | 120 | 120
Subjects
  Any Fatigue | 45 | 50 | 47 | 44 | 42 | 39 | 47
  Any Headache | 44 | 50 | 42 | 44 | 44 | 35 | 47
  Any Joint pain | 33 | 37 | 36 | 26 | 28 | 16 | 30
  Any Muscle aches | 54 | 52 | 59 | 49 | 48 | 42 | 55
  Any Shivering | 12 | 18 | 16 | 8 | 20 | 10 | 18
  Any Sweating | 15 | 20 | 15 | 11 | 14 | 10 | 11
  Any Fever | 2 | 5 | 6 | 3 | 8 | 2 | 2

9. Primary Outcome: Number of Subjects With Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s).
Time Frame: From Day 0 to Day 909
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 120 | 121 | 119 | 119 | 122 | 120 | 120
Subjects | 68 | 66 | 77 | 75 | 62 | 63 | 70

10. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as any occurrence of an unsolicited AE in a subject, regardless of intensity grade or relation to vaccination.
Time Frame: Within the 43-day (Days 0-42) post-vaccination periods
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 120 | 121 | 119 | 119 | 122 | 120 | 120
Subjects | 70 | 72 | 78 | 68 | 67 | 68 | 75

11. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A SAE was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as an occurrence of an SAE, regardless its relationship to vaccination.
Time Frame: From Day 0 to Day 909
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 120 | 121 | 119 | 119 | 122 | 120 | 120
Subjects | 12 | 14 | 11 | 9 | 11 | 15 | 12

12. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. Pre-vaccination for this outcome measure corresponds to Day 182. This outcome measure solely concerns subjects in the Naïve Placebo-A/turkey H5N1-Formulation 3 Group.
Time Frame: At Day 192
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 99
Subjects | 44

13. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey Virus Strain.
Description: HI antibody titers against the A/turkey virus strain were expressed as geometric mean titers (GMTs). This outcome measure solely concerns subjects in the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo and Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo groups.
Time Frame: At Days 182 and 192
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group
Number analyzed (Participants) | 95 | 92
Titers
  A/turkey, Day 182 (N=95,92) | 17.6 [13.1 to 23.6] | 12.2 [9.7 to 15.4]
  A/turkey, Day 192 (N=94,86) | 308.4 [231.1 to 411.5] | 374.4 [297.9 to 470.5]

14. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome measure solely concerns subjects in the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo and Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo groups.
Time Frame: At Days 182 and 192
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group
Number analyzed (Participants) | 95 | 92
Subjects
  A/turkey, Day 182 (N=95,92) | 30 | 25
  A/turkey, Day 192 (N=94,86) | 89 | 85

15. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome measure solely concerns subjects in the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo, Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo, and Naïve Placebo-A/turkey H5N1-Formulation 3 groups.
Time Frame: At Day 224
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 89 | 86 | 98
Subjects | 82 | 82 | 60

16. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: as for outcome 5
Time Frame: At Day 591
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group
Number analyzed (Participants) | 82 | 88 | 80 | 71
Subjects | 77 | 83 | 75 | 67

17. Secondary Outcome: Geometric Mean Fold Rise (GMFR) as Regards Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain
Description: GMFR was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the baseline reciprocal HI titer. Baseline for this outcome measure corresponds to Day 182. This outcome measure solely concerns subjects in the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo, Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo, and Naïve Placebo-A/turkey H5N1-Formulation 3 groups.
Time Frame: At Days 192 and 224
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 94 | 86 | 99
Fold increase
  A/turkey, Day 192 (N=94,86,99) | 17.8 [12.0 to 26.2] | 30.2 [22.2 to 41.2] | 4.0 [2.9 to 5.5]
  A/turkey, Day 224 (N=89,86,98) | 11.2 [7.8 to 16.3] | 17.2 [12.9 to 23.0] | 4.2 [3.0 to 5.7]

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) as Regards Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain
Description: GMFR was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the baseline reciprocal HI titer. Baseline for this outcome measure corresponds to Day 549. This outcome measure solely concerns subjects in the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 and Naïve Placebo-A/turkey H5N1-Formulation 3 groups.
Time Frame: At Day 559
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 83 | 88 | 80 | 72 | 81
Fold increase
  A/turkey, Day 559 (N=83,87,80,72,81) | 32.0 [21.9 to 46.8] | 32.0 [23.4 to 43.7] | 48.1 [34.6 to 66.9] | 30.1 [21.0 to 43.0] | 19.5 [13.4 to 28.4]
  A/turkey, Day 591 (N=82,88,80,71,81) | 26.7 [18.4 to 38.7] | 29.1 [21.3 to 39.9] | 35.2 [25.4 to 48.8] | 22.0 [15.8 to 30.7] | 14.8 [10.4 to 21.2]

19. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: as for outcome 1
Time Frame: At Day 591
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group
Number analyzed (Participants) | 82 | 88 | 80 | 71
Subjects | 69 | 80 | 70 | 61

20. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against the A/Turkey/Turkey/1/2005 (A/Turkey) Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. Pre-vaccination for this outcome measure corresponds to Day 182. This outcome measure solely concerns subjects in the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo, Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo, and Naïve Placebo-A/turkey H5N1-Formulation 3 groups.
Time Frame: At Day 224
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 89 | 86 | 98
Subjects | 64 | 75 | 42

21. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey) Strain.
Description: HI antibody titers against the A/turkey virus strain were expressed as geometric mean titers (GMTs). This outcome measure concerns solely the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo and Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo groups.
Time Frame: At Days 0, 182,192, 224, 549 and 729
Population: The analysis was performed on the Day 729 According-to-Protocol cohort for immunogenicity, i.e., all evaluable subjects with at least Day 182 and 192 or Day 549 and 559 haemagglutination inhibition (HI) titer results for the A/turkey/Turkey/1/05 virus), as well as with HI titers results available up to the Day 729 time point, for any virus strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group
Number analyzed (Participants) | 95 | 92
Titers
  A/turkey, Day 0 (N= 95,92) | 9.2 [7.4 to 11.4] | 6.6 [5.7 to 7.7]
  A/turkey, Day 182 (N=95,92) | 17.6 [13.1 to 23.6] | 12.2 [9.7 to 15.4]
  A/turkey, Day 192 (N=94,86) | 308.4 [231.1 to 411.5] | 374.4 [297.9 to 470.5]
  A/turkey, Day 224 (N=93,91) | 195.0 [146.7 to 259.1] | 213.7 [170.7 to 267.5]
  A/turkey, Day 549 (N=84,81) | 32.7 [24.4 to 43.6] | 28.7 [22.6 to 36.5]
  A/turkey, Day 729 (N=78,78) | 41.8 [32.1 to 54.4] | 31.2 [24.8 to 39.2]

22. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey) Strain.
Description: HI antibody titers against the A/turkey virus strain were expressed as geometric mean titers (GMTs). This outcome measure concerns solely the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4, and Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 groups.
Time Frame: At Days 0, 182, 549, 559, 591 and 729
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group
Number analyzed (Participants) | 90 | 96 | 99 | 89
Titers
  A/turkey, Day 0 (N=90,96,99,89) | 8.0 [6.6 to 9.8] | 7.1 [6.0 to 8.3] | 6.6 [5.7 to 7.6] | 6.9 [5.9 to 8.0]
  A/turkey, Day 182 (N=90,96,99,89) | 13.5 [10.3 to 17.8] | 10.8 [8.4 to 13.9] | 12.8 [10.0 to 16.4] | 13.7 [10.6 to 17.7]
  A/turkey, Day 549 (N=83,86,81,72) | 11.1 [8.8 to 14.1] | 8.4 [7.1 to 9.9] | 9.2 [7.6 to 11.2] | 11.4 [9.1 to 14.4]
  A/turkey, Day 559 (N=83,85,80,72) | 356.7 [265.9 to 478.5] | 266.4 [202.2 to 350.9] | 446.6 [336.0 to 593.7] | 343.9 [254.2 to 465.3]
  A/turkey, Day 591 (N=82,86,80,71) | 300.3 [225.6 to 399.7] | 242.4 [182.8 to 321.5] | 326.9 [241.6 to 442.2] | 254.4 [188.5 to 343.3]
  A/turkey, Day 729 (N=81,83,79,70) | 119.2 [95.3 to 149.0] | 96.6 [75.1 to 124.2] | 134.8 [106.4 to 170.9] | 105.6 [84.1 to 132.6]

23. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Turkey/Turkey/1/2005 (A/Turkey) Strain.
Description: HI antibody titers against the A/turkey virus strain were expressed as geometric mean titers (GMTs). This outcome measure concerns solely the Naïve Placebo-A/turkey H5N1-Formulation 3 Group.
Time Frame: At Days 0, 182, 192, 224, 549, 559, 591 and 729
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 99
Titers
  A/turkey, Day 0 (N=99) | 8.0 [6.6 to 9.7]
  A/turkey, Day 182 (N=99) | 10.6 [8.2 to 13.6]
  A/turkey, Day 192 (N=98) | 43.4 [32.5 to 58.0]
  A/turkey, Day 224 (N=98) | 43.7 [32.1 to 59.5]
  A/turkey, Day 549 (N=81) | 15.6 [12.0 to 20.2]
  A/turkey, Day 559 (N=80) | 314.4 [229.5 to 430.8]
  A/turkey, Day 591 (N=80) | 236.2 [172.3 to 323.8]
  A/turkey, Day 729 (N=80) | 98.1 [76.4 to 125.9]

24. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against the A/Turkey/Turkey/1/2005 Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome measure concerns solely the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo and Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo groups.
Time Frame: At Days 0, 182,192, 224, 549 and 729
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group
Number analyzed (Participants) | 95 | 92
Subjects
  A/turkey, Day 0 (N= 95,92) | 16 | 7
  A/turkey, Day 182 (N=95,92) | 30 | 25
  A/turkey, Day 192 (N=94,86) | 89 | 85
  A/turkey, Day 224 (N=93,91) | 86 | 87
  A/turkey, Day 549 (N=84,81) | 42 | 40
  A/turkey, Day 729 (N=78,78) | 47 | 49

25. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against the A/Turkey/Turkey/1/2005 Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome measure concerns solely the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4, and Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 groups.
Time Frame: At Days 0, 182, 549, 559, 591 and 729
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group
Number analyzed (Participants) | 90 | 96 | 99 | 89
Subjects
  A/turkey, Day 0 (N=90,96,99,89) | 11 | 8 | 8 | 6
  A/turkey, Day 182 (N=90,96,99,89) | 25 | 20 | 28 | 31
  A/turkey, Day 549 (N=83,86,81,72) | 15 | 8 | 10 | 13
  A/turkey, Day 559 (N=83,85,80,72) | 79 | 81 | 77 | 69
  A/turkey, Day 591 (N=82,86,80,71) | 77 | 82 | 75 | 67
  A/turkey, Day 729 (N=81,83,79,70) | 75 | 73 | 71 | 66

26. Secondary Outcome: Number of Subjects Seroprotected for HI Antibodies Against the A/Turkey/Turkey/1/2005 Virus Strain
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody titers against the A/turkey virus strain greater than or equal to (≥) 1:40. This outcome measure concerns solely the Naïve Placebo-A/turkey H5N1-Formulation 3 Group.
Time Frame: At Days 0, 182, 192, 224, 549, 559, 591 and 729
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 99
Subjects
  A/turkey, Day 0 (N=99) | 8
  A/turkey, Day 182 (N=99) | 23
  A/turkey, Day 192 (N=98) | 63
  A/turkey, Day 224 (N=98) | 59
  A/turkey, Day 549 (N=81) | 21
  A/turkey, Day 559 (N=80) | 76
  A/turkey, Day 591 (N=80) | 73
  A/turkey, Day 729 (N=80) | 70

27. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Indonesia/5/05 (A/Indo) Virus Strain.
Description: HI antibody titers against the A/Indo virus strain were expressed as geometric mean titers (GMTs). This outcome measure solely concerns the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo and Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo groups.
Time Frame: At Days 0, 10, 42, 182 and 549
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group
Number analyzed (Participants) | 95 | 92
Titers
  A/Indo, Day 0 (N=95,92) | 6.7 [5.7 to 7.9] | 5.9 [5.4 to 6.5]
  A/Indo, Day 10 (N=95,92) | 32.3 [23.5 to 44.4] | 30.7 [23.4 to 40.4]
  A/Indo, Day 42 (N=93,88) | 44.1 [32.4 to 59.9] | 44.8 [34.7 to 57.9]
  A/Indo, Day 182 (N=95,92) | 22.4 [16.7 to 30.0] | 15.7 [12.3 to 20.0]
  A/Indo, Day 549 (N=84,81) | 24.0 [17.3 to 33.2] | 22.7 [17.6 to 29.4]

28. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against the A/Indonesia/5/05 (A/Indo) Virus Strain.
Description: HI antibody titers against the A/Indo virus strain were expressed as geometric mean titers (GMTs). This outcome measure solely concerns the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2, and Naïve Placebo-A/turkey H5N1-Formulation 3 groups.
Time Frame: At Days 0, 10, 42, 182, 549 and 559
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 90 | 96 | 99 | 89 | 99
Titers
  A/Indo, Day 0 (N=90,96,99,89,99) | 5.9 [5.4 to 6.5] | 5.7 [5.3 to 6.2] | 5.7 [5.1 to 6.3] | 5.6 [5.1 to 6.1] | 5.9 [5.3 to 6.5]
  A/Indo, Day 10 (N=89,95,98,87,97) | 27.0 [19.4 to 37.6] | 17.2 [13.2 to 22.3] | 31.7 [24.2 to 41.4] | 26.2 [19.2 to 35.8] | 6.3 [5.6 to 7.1]
  A/Indo, Day 42 (N=87,94,96,87,97) | 37.5 [27.9 to 50.4] | 27.3 [21.0 to 35.4] | 45.7 [35.0 to 59.7] | 36.6 [27.1 to 49.5] | 6.2 [5.5 to 7.0]
  A/Indo, Day 182 (N=90,96,99,89,99) | 16.4 [12.5 to 21.6] | 13.7 [10.8 to 17.5] | 17.8 [14.0 to 22.6] | 16.2 [12.5 to 21.1] | 6.7 [5.8 to 7.7]
  A/Indo, Day 549 (N=83,86,81,72,81) | 8.1 [6.6 to 10.0] | 7.9 [6.7 to 9.4] | 7.8 [6.5 to 9.3] | 9.2 [7.4 to 11.3] | 6.2 [5.5 to 6.9]
  A/Indo, Day 559 (N=83,85,81,72,80) | 304.3 [232.4 to 398.5] | 231.9 [177.1 to 303.5] | 376.6 [285.2 to 497.2] | 289.2 [215.8 to 387.7] | 113.1 [82.4 to 155.3]

29. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/Indonesia/5/05 (A/Indo) Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody reciprocal titers against the A/Indo virus strain greater than or equal to (≥) 1:40. This outcome measure solely concerns the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo and Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo groups.
Time Frame: At Day 0, Day 10, Day 42, Day 182 and Day 549
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 95 | 92 | 99
Subjects
  A/Indo, Day 0 (N=95,92) | 6 | 6.7 | 2
  A/Indo, Day 10 (N=95,92) | 50 | 32.3 | 4
  A/Indo, Day 42 (N=93,88) | 57 | 44.1 | 3
  A/Indo, Day 182 (N=95,92) | 42 | 22.4 | 9
  A/Indo, Day 549 (N=84,81) | 38 | 24.0 | 2

30. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against A/Indonesia/5/05 (A/Indo) Virus Strain.
Description: A seroprotected subject was defined as a vaccinated subject with HI antibody reciprocal titers against the A/Indo virus strain greater than or equal to (≥) 1:40. This outcome measure solely concerns the Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2, and Naïve Placebo-A/turkey H5N1-Formulation 3 groups.
Time Frame: At Day 0, Day 10, Day 42, Day 182, Day 549, and Day 559
Population: as for outcome 21
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 90 | 96 | 99 | 89 | 99
Subjects
  A/Indo, Day 0 (N=90,96,99,89,99) | 1 | 0 | 3 | 2 | 2
  A/Indo, Day 10 (N=89,95,98,87,97) | 41 | 36 | 56 | 44 | 4
  A/Indo, Day 42 (N=87,94,96,87,97) | 50 | 51 | 68 | 53 | 3
  A/Indo, Day 182 (N=90,96,99,89,99) | 28 | 29 | 35 | 32 | 9
  A/Indo, Day 549 (N=83,86,81,72,81) | 9 | 9 | 7 | 11 | 2
  A/Indo, Day 559 (N=83,85,81,72,80) | 79 | 80 | 77 | 68 | 68

31. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against the A/Indo Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. Pre-vaccination for this outcome measure corresponds to Day 0.
  This outcome measure only concerns the Pumarix Primed-A/turkey H5N1-Formulation 1-Placebo, Pumarix Primed-A/turkey H5N1-Formulation 2-Placebo, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 3, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 1, Pumarix Primed-Placebo-A/turkey H5N1-Formulation 4 and Pumarix Primed-Placebo-A/turkey H5N1-Formulation 2 groups.
Time Frame: At Days 10 and 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Pumarix Primed-A/Turkey H5N1-Formulation 1-Placebo Group | Pumarix Primed-A/Turkey H5N1-Formulation 2-Placebo Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 3 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 1 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 4 Group | Pumarix Primed-Placebo-A/Turkey H5N1-Formulation 2 Group
Number analyzed (Participants) | 95 | 92 | 89 | 97 | 98 | 87
Subjects
  A/Indo, Day 10 (N=95,92,89,97,98,87) | 42 | 50 | 38 | 33 | 52 | 40
  A/Indo, Day 42 (N=93,88,87,96,96,87) | 50 | 61 | 49 | 51 | 64 | 51

32. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against the A/Indo Virus Strain.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer less than (<) 1:10 and a post-vaccination reciprocal titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. This outcome measure only concerns the Naïve Placebo-A/turkey H5N1-Formulation 3 Group, for whom the pre-vaccination time point corresponds to the Day 192 time point.
Time Frame: At Days 192 and 224
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Number analyzed (Participants) | 47
Subjects
  A/Indo, Day 192 | 8
  A/Indo, Day 224 | 3

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs): From Day 0 to Day 909; Solicited local and general symptoms: During the 7-day (Days 0-6) post vaccination periods; Unsolicited adverse events: During the 43-day (Days 0-42) post vaccination periods.
Groups:
- Naïve Placebo-A/Turkey H5N1-Formulation 3 Group: Healthy subjects aged 18 years of age or older at the time of vaccination received one dose of placebo (phosphate buffered saline, PBS) at Day 0 followed by two doses of A/turkey H5N1 vaccine formulation 3, one dose administered at Day 182 and the other at Day 549. Placebo vaccine and one dose of A/turkey H5N1 vaccine (Day 549) was administered intramuscularly in the deltoid region of the non-dominant arm while the other dose of A/turkey H5N1 vaccine (Day 182) was administered intramuscularly in the deltoid region of the dominant arm.
Arm/Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F1-Placebo Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F2-Placebo Group | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group
Serious Adverse Events (participants affected / at risk) | 12/120 | 14/121 | 11/119 | 9/119 | 11/122 | 15/120 | 12/120
Other Adverse Events (participants affected / at risk) | 106/120 | 109/121 | 106/119 | 103/119 | 106/122 | 101/120 | 106/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F1-Placebo Group (N=120) | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F2-Placebo Group (N=121) | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group (N=119) | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group (N=119) | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group (N=122) | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group (N=120) | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group (N=120)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endocarditis noninfective (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F1-Placebo Group (N=120) | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F2-Placebo Group (N=121) | A/Indonesia Primed-A/Turkey Influenza (H5N1)-F3-Placebo Group (N=119) | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F1-Group (N=119) | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F4-Group (N=122) | A/Indonesia Primed-Placebo-A/Turkey Influenza (H5N1)-F2-Group (N=120) | Naïve Placebo-A/Turkey H5N1-Formulation 3 Group (N=120)
Pain (General disorders) | 98 | 100 | 101 | 93 | 102 | 90 | 95
Redness (General disorders) | 8 | 4 | 12 | 9 | 14 | 4 | 8
Swelling (General disorders) | 6 | 7 | 15 | 4 | 16 | 9 | 11
Fatigue (General disorders) | 45 | 50 | 47 | 44 | 42 | 39 | 47
Headache (General disorders) | 44 | 50 | 47 | 44 | 44 | 35 | 47
Joint pain (General disorders) | 33 | 37 | 36 | 44 | 42 | 39 | 30
Muscle aches (General disorders) | 54 | 52 | 59 | 49 | 48 | 42 | 55
Shivering (General disorders) | 12 | 18 | 16 | 8 | 20 | 10 | 18
Sweating (General disorders) | 15 | 20 | 15 | 11 | 14 | 10 | 18
Fever (General disorders) | 2 | 5 | 6 | 3 | 8 | 2 | 2
Nasopharyngitis (Infections and infestations) | 15 | 9 | 9 | 14 | 12 | 11 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 9 | 12 | 1 | 10 | 11
Headache (Nervous system disorders) | 8 | 11 | 4 | 6 | 6 | 10 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 6 | 5 | 4 | 5 | 5
Nausea (Gastrointestinal disorders) | 2 | 2 | 10 | 6 | 3 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 4 | 8 | 4 | 5 | 7
Upper respiratory tract infection (Infections and infestations) | 7 | 5 | 6 | 3 | 6 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.